CLINICAL TRIAL: NCT03182959
Title: A Phase 0 Study Evaluating the Systemic Bioavailability and Pharmacodynamic Effects of Avmacol® in the Oral Mucosa of Patients Following Curative Treatment for Tobacco-related Head and Neck Cancer
Brief Title: Broccoli Sprout Extract in Preventing Recurrence in Patients With Tobacco-Related Head and Neck Squamous Cell Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 1612032762; 5P50CA097190 (NIH)
Record Dates: First submitted 2017-05-18; First posted 2017-06-09 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: HNSCC; Head and Neck Cancer; Head and Neck Squamous Cell Carcinoma; Tobacco-Related Carcinoma; Carcinoma in Situ; Dysplasia; Hyperplasia; Premalignant Lesion
Keywords: Nrf2 pathway; Oral mucosa; HNSCC; Head and Neck Cancer; Head and Neck Squamous Cell Carcinoma; Avmacol; Tobacco-related Head and Neck Cancer; broccoli sprout powder; broccoli seed extract powder
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms; Carcinoma in Situ; Hyperplasia

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive either 50 mg glucoraphanin (GR) in Cycle 1 and 100 mg GR in cycle 2, or 100 mg GR in Cycle 1 and 50 mg GR in Cycle 2, but all participants will receive both doses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lower dose, higher dose (Experimental): During the first cycle, the patient will self-administer Avmacol® (70 μmol/day SF equivalent) starting on the evening of Day 1 of the cycle. Participants will self-administer four tablets of Avmacol® every evening, ideally between 4 pm and 8 pm, through the evening of Day 28. Participants will record the date and time of each Avmacol® administration on the provided diary.
  During the second cycle, the patient will self-administer Avmacol® (140 μmol/day SF equivalent) starting on the evening of Day 1 of the cycle. Participants will self-administer eight tablets of Avmacol® every evening, ideally between 4 pm and 8 pm, through the evening of Day 28. Participants will record the date and time of each Avmacol® administration on the provided diary.
  Interventions: Drug: Avmacol®
- Higher dose, lower dose (Experimental): During the first cycle, the patient will self-administer Avmacol® (140 μmol/day SF equivalent) starting on the evening of Day 1 of the cycle. Participants will self-administer eight tablets of Avmacol® every evening, ideally between 4 pm and 8 pm, through the evening of Day 28. Participants will record the date and time of each Avmacol® administration on the provided diary.
  During the second cycle, the patient will self-administer Avmacol® (70 μmol/day SF equivalent) starting on the evening of Day 1 of the cycle. Participants will self-administer four tablets of Avmacol® every evening, ideally between 4 pm and 8 pm, through the evening of Day 28. Participants will record the date and time of each Avmacol® administration on the provided diary.
  Interventions: Drug: Avmacol®

INTERVENTIONS:
Drug: Avmacol® — Avmacol® tablets
  Other Names: Broccoli Sprout Extract

SUMMARY:
This study is being done to see whether Avmacol®, a dietary supplement made from broccoli sprout and seed extract powder, induces changes in inner cheek cells that may be protective against environmental toxins such as tobacco.

There are three main goals of the study:

1. To learn whether the dietary supplement, Avmacol®, can stimulate cheek cells to repair damage from environmental toxins;
2. to learn how the body metabolizes Avmacol®, by measuring its byproducts in the participant's urine and blood;
3. to learn whether the immune system can be stimulated by Avmacol®, by studying the natural killer cells and T cells in the participant's blood.

DETAILED DESCRIPTION:
This study hypothesizes that nuclear factor erythroid 2-related factor 2 (NRF2) pathway activation in oral epithelium can be induced by administering Avmacol® to patients curatively treated for a first tobacco-related HNSCC.

The aim of this Phase 0 clinical study is to determine the oral bioavailability of sulforaphane in the commercially available dietary supplement, Avmacol®, and to determine the level of pharmacodynamic upregulation of NRF2 target gene transcripts that occurs in the oral epithelium of patients who have completed curative treatment for tobacco-related HNSCC, including high grade dysplasia, carcinoma in situ, or invasive carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have completed curative-intent therapy (including surgery, radiation, and/or chemotherapy) for a first tobacco-related oral premalignant lesion (OPL) or HNSCC of any stage (eligible lesions include high grade dysplasia; carcinoma in situ; or stage I-IVa HNSCC).
* Primary site may include oral cavity, pharynx, or larynx. Oropharynx primaries must be human papillomavirus (HPV) negative as defined by routine p16 IHC at the local site.
* Patients may be enrolled between 3 months and 5 years AFTER completion of curative-intent therapy (including surgery, radiotherapy, and/or chemotherapy).
* Patients may have untreated OPLs (i.e., hyperplasia, dysplasia, carcinoma in situ) at the time of study entry, provided the index OPL or HNSCC was definitively treated.
* Patients must have a Karnofsky Performance Status of 80% or higher or an Eastern Cooperative Oncology Group (ECOG) of 0-1
* Current and former tobacco users are eligible.
* Able to perform written, informed consent.
* Women of childbearing potential (WCBP) must have a negative urine pregnancy test within 7 Days prior to the first study intervention.
* WCBP and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study and for the duration of study participation.

Exclusion Criteria:

* Patient has a history of another malignancy within 2 years prior to starting study treatment, except for excised and cured carcinoma-in-situ of breast or cervix; non-melanomatous skin cancer; T1-2, N0, M0 differentiated thyroid carcinoma either resected or under active surveillance; superficial bladder cancer; T1a or T1b prostate cancer comprising < 5% of resected tissue with normal prostate specific antigen (PSA) since resection, or status post external beam radiation or brachytherapy with normal PSA since radiation.
* Primary oropharyngeal HNSCC which is HPV (+) as defined by p16 immunohistochemistry.
* Participants with acute intercurrent illness or those who had major surgery within the preceding 4 weeks unless they have fully recovered.
* Participants who have a positive pregnancy test, are pregnant, or breast feeding.
* Patients who are not practicing adequate contraception are ineligible if they are of child bearing potential.
* Patients currently using anti-neoplastic or anti-tumor agents, including chemotherapy, radiation therapy, immunotherapy, and hormonal anticancer therapy.
* Chronic anticoagulation with warfarin. Patients on low molecular weight heparin or fondaparinux may be enrolled.
* Use of chronic prescribed medications which are potent inducers or inhibitors of CYP3A4
* Chronic use of steroids at immunosuppressive doses.
* History of severe food intolerance to broccoli.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2021-01-19 (Actual)

PRIMARY OUTCOMES:
Determine whether Avmacol® results in acute and/or sustained induction of NRF2 target gene transcripts in the oral mucosa of patients who have been curatively treated for a tobacco-related HNSCC. | 4 months
  Quantitative changes in NRF2 target gene transcripts (i.e. NAD(P)H Quinone Dehydrogenase 1 [NQO1] and GCLC) in buccal cytobrush by quantitative polymerase chain reaction (qPCR) according to a linear mixed model framework.

SECONDARY OUTCOMES:
Determine whether NRF2 target protein expression is upregulated by Avmacol® in the oral mucosa. | 4 months
  Change in NRF2 target proteins in buccal punch biopsies by immunoblotting.
Evaluate for a dose-response relationship between Avmacol® dose and quantitative change in candidate NRF2 pathway biomarkers in oral mucosa. | 4 months
  Acute change in NRF2 target gene transcripts, as compared to baseline, between the two doses of Avmacol®.
Evaluate oral mucosa for quantitative modulation of NRF2-independent biomarkers of sulforaphane (SF) chemopreventive efficacy, as defined in parallel preclinical models. | 4 months
  Change in NRF2-independent proteins by immunoblotting, eg. STAT3, phospho-STAT3 (pSTAT3).
Evaluate biomarkers of Avmacol® activity in PBMCs gene expression | 4 months
  Alterations in Peripheral Blood Mononuclear Cells (PBMC) gene expression patterns
Evaluate biomarkers of Avmacol® activity in PBMCs flow cytometry | 4 months
  Alterations in Peripheral Blood Mononuclear Cells (PBMC) immune cell sub-populations
Evaluate biomarkers of Avmacol® activity in PBMCs functional assays of T cells and NK cells | 4 months
  Alterations in Peripheral Blood Mononuclear Cells (PBMC) Tcell/ Natural Killer (NK) cell function
Evaluate cytokine biomarkers of Avmacol® activity in serum, including CXCL8, Interleukin 8 (IL8). | 4 months
  Change in serum cytokine levels, as determined by multiplexed bead-based cytokine assays.
Measurement of serum albumin-bound SF using isotope dilution mass spectrometry. | 4 months
  Sulforaphane metabolites will be assessed in overnight urine collected following the first dose of each cycle. The steady state concentration of broccoli seed preparations will be characterized by measuring albumin-bound sulforaphane in serum collected on the last day of each cycle. This assay represents an integrated measure of sulforaphane exposure, which will be correlated with biomarker modulation by means of repeated measures analysis of covariance.
Measure urinary metabolites of SF during administration of two doses of Avmacol®. | 4 months
  Measurement of urinary metabolites of SF using isotope dilution mass spectrometry.
Description of safety profile in accordance with NCI CTCAE v.4. | 4 months
  Patients will receive a diary for daily logging of adverse events. This will tabulated by Avmacol dose and type and grade of adverse events. The mean frequency and grade of events will be calculated by dose, and between-dose differences compared by means of mixed effects analysis of covariance.
Description of the proportion of patients with HNSCC primary tumors harboring genomic alteration of NRF2. | 4 months
  Describe the genetic profile of NRF2 within the index HNSCC primary tumor in the target population.
  Archived tumor specimens from the index tobacco-related head and neck squamous cell carcinoma will be collected. Tumor specimens analyzed for genomic alterations in NRF2 and related genes. The frequency of genomic alterations will be characterized.
Description of the proportion of patients with HNSCC primary tumors harboring genomic alteration of NRF2 related genes. | 4 months
  Describe the genetic profile of other related genes within the index HNSCC primary tumor in the target population.
  Archived tumor specimens from the index tobacco-related head and neck squamous cell carcinoma will be collected. Tumor specimens analyzed for genomic alterations in NRF2 and related genes. The frequency of genomic alterations will be characterized.

CONTACTS AND LOCATIONS:
Overall Officials: Julie E. Bauman, MD, MPH, Principal Investigator — The University of Arizona
Locations (1):
- The University of Arizona Cancer Center, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided